CLINICAL TRIAL: NCT00801476
Title: A Prospective Cohort Study to Evaluate the Impact of Preoperative Breast Magnetic Resonance Imaging (MRI) on Surgical Decision-Making in Young Patients With Breast Cancer
Brief Title: Pre-operative Magnetic Resonance Imaging (MRI) in Young Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Responsible Party: Dr. Nicole Hodgson, Juravinski Cancer Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MRI REB 07-458
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2009-11

CONDITIONS: Breast Cancer; Magnetic Resonance Imaging; Preoperative MRI
Keywords: Breast Cancer; Magnetic Resonance Imaging; Preoperative MRI
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Pre-operative bilateral breast MRI — After the standard mammogram and ultrasound testing, the surgeon is asked which surgical procedure they feel is appropriate for the patient. A bilateral breast MRI is then performed prior to surgery. The surgeon is again asked which surgery they feel is appropriate based on the new information provided by the MRI. The study is trying to see if this pre-operative breast MRI helps define the tumour leading to a better first surgical decision.
  Other Names: No "Other names" for this study

SUMMARY:
Young women with breast cancer have an increased breast tissue density and conventional imaging tests such as mammography and breast ultrasound are less sensitive and specific for detecting breast cancer than in older breast cancer patients. Breast MRI is an emerging tool that has been proven to improve the ability to identify breast cancers by determining the extent of disease and also detect multifocal, multicentric and bilateral breast cancers. To date, the role of pre-operative breast MRI is not clearly defined. The investigators are proposing a study to evaluate the impact of preoperative breast MRI on surgical decision-making in breast cancer patients <= 50 years. This may lead to improved characterization of breast cancers in these younger patients that may ultimately result in lower local recurrence rates in the future. The additional information attained through the breast MRI may also guide the use of radiation, chemotherapy and/or hormonal therapy in these patients.

DETAILED DESCRIPTION:
Inclusion Criteria:

* female aged ≤ 50
* histologically proven invasive breast cancer

Exclusion Criteria:

* Is not considered a surgical candidate
* Has had prior breast cancer surgery or an excisional biopsy of the newly diagnosed lesion
* Has a contraindication to undergoing breast MRI
* Has inflammatory breast cancer according to the standard clinical definition
* Has locally advanced breast cancer according to the standard clinical definition
* Patient is pregnant
* Has a psychiatric or addictive disorder that would preclude obtaining informed consent or adherence to the protocol

ELIGIBILITY:
Inclusion Criteria:

* Female aged <= 50 years
* Histological proof of invasive breast cancer via fine needle aspiration or core needle biopsy
* Premenopausal

Exclusion Criteria:

* Patient not considered an appropriate surgical candidate; i.e., patient is not well enough to have breast cancer surgery
* Patient has had prior breast cancer surgery or an excisional biopsy of the newly diagnosed cancer
* Patient has a contraindication to undergoing breast MRI (i.e., pacemaker, neurodefibrillator, metallic foreign bodies, etc.)
* Patient has inflammatory breast cancer according to the standard clinical definition. This is a type of breast cancer in which there is evidence of erythema and/or edema. The skin of the breast may also have changes of peau d'orange.
* Patient has locally advanced breast cancer according to the standard clinical definition.
* Patient is pregnant
* Patient has a psychiatric or addictive disorder that would preclude them from obtaining informed consent.

Max Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-12 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Does pre-operative magnetic resonance imaging (MRI) effect surgical management in young women with breast cancer | 3 months

SECONDARY OUTCOMES:
Proportion of patients requiring a second surgery due to positive tumour margins. | 3 months
Incidence of multifocal or multicentric or bilateral breast cancer found on MRI | After surgery
The correlation between MRI tumour size and the pathologic tumour size after surgery. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Hodgson, MD, Principal Investigator — Juravinski Cancer Centre; Som D Mukherjee, MD, Principal Investigator — Juravinski Cancer Centre
Locations (2):
- Canada (2):
  - St. Josephs' Healthcare, Hamilton, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario